CLINICAL TRIAL: NCT03641833
Title: Identification of Factors Causing Postoperative Cognitive Dysfunction in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass (CPB)
Brief Title: Identification of Factors Causing Postoperative Cognitive Dysfunction in Patients Undergoing Cardiac Surgery With CPB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rasa Bukauskiene (Other)
Responsible Party: Sponsor-Investigator, Rasa Bukauskiene, Physician anaesthesiologist, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: POCD-1
Record Dates: First submitted 2018-07-15; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: cardiac; surgery; postoperative cognitive dysfunction; bypass; brain biomarkers; transcranial Doppler
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood sample for brain biomarkers — Transcranial Doppler will be performed to evaluate a.cerebri media blood flow speed during surgery.
  Other Names: device

SUMMARY:
The incidence of cognitive decline occurs in 53% of patients after cardiac surgery. Causes of POCD can be various: age, duration of cardiac bypass, medicaments and many others. The aim of this study is to determine factors causing postoperative cognitive dysfunction (POCD) and to identify which of them are most important

DETAILED DESCRIPTION:
Prospective case-control study included patients undergoing cardiac at Clinic of Cardiac, Vascular and Thoracic Surgery, Lithuanian University of Health Sciences. Inclusion criteria is: 1) cardiac output > 35%; 2) no agents affecting central nervous system; 3) no neuropathology; 5) no multiple organ dysfunction. Patients will have to perform mini mental state examination (MMSE), Trial making, addenbrooke tests before and 7 days after surgery. Brain biomarkers glial fibrillary acid protein (GFAP) and neurofilaments will be taken after induction, 24 and 48 hours after surgery. Transcranial Doppler will be performed to evaluate a.cerebri media blood flow speed during surgery.

After these test, the investigators are going to examine data about patient and operation, recognize factors causing POCD and identify the most important of them.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass grafting or/and heart valve surgery;
* Patients age>18years
* Cardiac output >35%

Exclusion Criteria:

* Patient disagreement;
* Diseases causing cognitive dysfunction;
* Multi organic deficiency;
* Agents affecting central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study include patients undergoing cardiac at Clinic of Cardiac, Vascular and Thoracic Surgery, Lithuanian University of Health Sciences
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Brain blood flow speed changes during surgery and correlation with POCD | 3 years
  Transcranial Doppler will be performed to evaluate a.cerebri media blood flow speed during surgery using the 2MHz TCD ultrasound transducer over the temporal area. By adjusting the probe the curve of arteria will appear. Target measurement- mean flow velocity (MFV is measured in cm/s).

SECONDARY OUTCOMES:
Brain biomarker GFAP concentration chances before and after surgery and correlation with POCD. | 3 years
  Blood sample for brain biomarkers GFAP will be taken after induction, 24 and 48 hours after surgery. GFAP concentration in blood serum is measured in ng/ml
Brain biomarker neurofilaments concentration chances before and after surgery and correlation with POCD. | 3 years
  Blood sample for brain biomarker neurofilaments will be taken after induction, 24 and 48 hours after surgery. GFAP concentration in blood serum is measured in pg/ml

OTHER OUTCOMES:
Determine factors causing POCD | 3 years
  Patients will complete questionares: mini mental state examination (MMSE), Trial making and addenbrooke test one day before and 10 days after the surgery. We are going to compare change in tests results after surgery and find correlation with brain biomarkers and blood flow speed during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Outside US/Canada/Australia, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided